CLINICAL TRIAL: NCT06411678
Title: Application of 68GA-labeled CD73 Targeting Probe PET/CT Imaging in the Diagnosis of Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-CD73
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68GA-DOTA-dPNE (Experimental): Each patient receive a single intravenous injection of 68GA-DOTA-dPNE 0.5-0.6 mci/kg and undergo PET/CT
  Interventions: Drug: 68GA-DOTA-dPNE

INTERVENTIONS:
Drug: 68GA-DOTA-dPNE — Patients with breast cancer receive intravenously 68GA-DOTA-dPNE followed by PET/CT after 40min of injection

SUMMARY:
The investigators plan to conduct a 68Ga-DOTA-dPNE PET/CT imaging study in breast cancer patients to observe the binding of the tracer to tumor lesions and evaluate CD73 expression. As part of the study design, a subset of patients will initially undergo dynamic PET/CT imaging to evaluate the safety profile and pharmacokinetic distribution of the radiotracer in vivo. Subsequently, static PET/CT imaging will be performed on additional patients to assess the diagnostic effectiveness of 68Ga-DOTA-dPNE. Imaging results will be correlated with relevant clinical indicators to evaluate the potential of this tracer in diagnosing breast cancer, guiding therapeutic decisions, and predicting responses to targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged ≥18 years with an expected survival of at least 12 weeks No prior radiotherapy or chemotherapy; surgery or biopsy is feasible for pathological diagnosis At least one measurable target lesion as defined by RECIST v1.1 Able to provide written informed consent and comply with follow-up requirements

Exclusion Criteria:

Severe hepatic or renal dysfunction Pregnant, breastfeeding, planning to become pregnant, or planning to have children during the study period; women of childbearing potential must use effective contraception during the study Unable to lie flat for 30 minutes History of claustrophobia or other psychiatric disorders Any other condition deemed unsuitable for participation by the investigator Refusal to participate in the clinical study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The evaluation of diagnostic performance of 68Ga-DOTA-dPNE PET in breast cancer | through study completion, an average of 1 year
  Patients with histologically proven breast cancer will be prospectively recruited in this study. They will receive 68Ga-DOTA-dPNE and 18F-FDG. The detection rates of lesions, bones and lymph nodes (visual) were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Xianzhong ZHANG, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- PUMCH, Dongcheng, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No